CLINICAL TRIAL: NCT01162577
Title: Oklahoma Weight Concerns Quitline: a Randomized Cessation Trial
Acronym: OKRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consumer Wellness Solutions (Industry)
Collaborators: Oklahoma Tobacco Settlement Endowment Trust (TSET) (Unknown)
Responsible Party: Terry Bush PhD, Associate Investigator, Free & Clear, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Smoking
Keywords: Weight; Smoking; Quitline
MeSH Terms: conditions — Smoking; Body Weight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervetion (Experimental): The intervention group received the 5 standard tobacco calls plus 3 weight calls with a weight coach to address weight concerns related to quitting smoking
  Interventions: Behavioral: Weight Concerns
- Control (No Intervention): Participants in this arm received only the 5 standard tobacco calls

INTERVENTIONS:
Behavioral: Weight Concerns — Standard Quitline plus weight coaching
  Other Names: Standard Quitline
  Arms: Intervetion

SUMMARY:
The purpose of the "Weigh2Quit" study was to test in a randomized trial, a "weight concerns" intervention designed to reduce weight concerns that might impact cessation, increase physical activity and adherence to tobacco treatment, increase confidence in quitting, improve tobacco quit rates and decrease weight gain post-quit.

DETAILED DESCRIPTION:
Smoking and obesity are the two biggest contributors to preventable morbidity and mortality. They are usually thought of independently, but for many people are inter-related. Cessation-related weight gain and concerns about weight gain are common and negatively impact cessation efforts.

Between March 2008 and November 2008 smokers who called the OKHL were screened for the presence of weight concerns and asked if they would be interested in a study offering the chance to speak with a weight coach (WC). Interested individuals were transferred to a specially trained Quit Coach (QC) who provided informed verbal consent, collected additional baseline data, obtained a second verbal consent to be randomized and were then randomized using a pre-programmed automated randomization procedure. Groups were randomly assigned in blocks of 20 so that after every 20th person randomized, the cells would be balanced. Individuals were randomized into either the control group to receive the standard quitline only (the OKHL 5-call program), or into the intervention group to receive standard care with integrated weight content plus three calls with a weight coach. All participants were offered a total of five tobacco cessations calls, access to Web Coach, tailored emails with quitting tips, access to the inbound support line, mailed quit guides, and nicotine replacement therapy (NRT) for cessation as appropriate. For the intervention group, QCs and WCs integrated weight concerns topics and components of the tobacco treatments into their calls with the primary goal of smoking cessation. A 6-month follow-up survey was conducted by the Oklahoma Tobacco Research Center, University of Oklahoma Health Sciences Center to compare outcomes between intervention and control conditions. The primary outcome was the 30-day quit rate. Secondary outcomes were:

90 day abstinence, adherence to tobacco treatment, confidence in quitting or staying quit, confidence in controlling weight gain after quitting, change in physical activity, participant satisfaction, change in weight concerns, change in weight by quit outcomes

We hypothesized that relative to controls, the 'Weight2Quit' intervention would:

1. increase cessation without excessive weight gain
2. increase satisfaction with the OKHL
3. increase call completion rate
4. reduce weight concerns, and
5. increase confidence in quitting without weight gain THE STANDARD QUITLINE CESSATION PROGRAM The 5 proactive calls provided to participants in the multiple call programs are scheduled by mutual agreement between each participant and his or her Quit Coach. The aim is to set a quit date within 15 days, schedule calls around that quit date, and complete all calls within three months of enrollment.

THE WEIGH2QUIT INTERVENTION The intervention was modeled on evidence-based methods to address maladaptive weight gain concerns that negatively impact quitting (Perkins, 2001). In this study, we adapted the original intensive, in-person group intervention described by Perkins for delivery via a telephone-based quitline. Participants randomized to the Weigh2Quit intervention were offered the standard OKHL cessation program (with integrated weight concerns content) plus 3 additional calls with a weight coach and specialized support materials. The mailed materials included a description of the rationale of the new program, educational information and worksheets (e.g. self-monitoring forms for tracking maladaptive thoughts about weight and body image and tracking alternative thoughts). Intervention counseling calls were designed to increase smoking cessation and

ELIGIBILITY:
Inclusion Criteria:

* Individuals were eligible for the study if they were age 18 or older, smoked at least 5 cigarettes per day, were willing to quit within 30 days from enrollment in the Helpline, were not pregnant or nursing, agreed to be in the study and randomized, agreed to the follow-up interview, provided a workable phone number with a secondary back-up number, had a BMI of at least 23 and reported having significant concerns about gaining weight with quitting.

Exclusion Criteria:

* Individuals were not eligible for the study if they had a BMI lower than 23 or were pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
30 day abstinence | 6 months
  No smoking in the past 30 days

SECONDARY OUTCOMES:
Change in weight | 6 months
  Change in weight (pounds)between baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Terry Bush, PhD, Principal Investigator — Free & Clear, Inc.
Locations (1):
- Free & Clear, Seattle, Washington, United States

REFERENCES:
- [Result] Bush T, Levine MD, Deprey M, Cerutti B, Zbikowski SM, McAfee T, Mahoney L, Beebe L. Prevalence of Weight Concerns and Obesity Among Smokers Calling a Quitline. J Smok Cessat. 2008 Dec 1;4(5):74-78. doi: 10.1375/jsc.4.2.74. PMID 20548969
- [Derived] Bush T, Levine MD, Beebe LA, Cerutti B, Deprey M, McAfee T, Boeckman L, Zbikowski S. Addressing weight gain in smoking cessation treatment: a randomized controlled trial. Am J Health Promot. 2012 Nov-Dec;27(2):94-102. doi: 10.4278/ajhp.110603-QUAN-238. PMID 23113779